CLINICAL TRIAL: NCT05603325
Title: Facilitating the Use of Patient Experience Feedback to Improve Mental Health Inpatient Services - a Feasibility and Acceptability Study.
Brief Title: Using Patient Feedback in Mental Health Services
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1-089-22
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Patient Participation
Keywords: mental health; patient feedback; person centered practice development
MeSH Terms: conditions — Patient Participation; Psychological Well-Being | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient participants: Current inpatients within the acute mental health ward in which the study is taking place.
  Interventions: Other: Interview
- Staff participants: Staff working within the acute mental health ward in which the study is taking place including nursing, mental, occupational therapy, estate and management team members
  Interventions: Other: Person Centered Practice

INTERVENTIONS:
Other: Person Centered Practice — Staff will be asked to:
  * Complete two surveys on two occasions, once before the intervention sessions and once following the last session. The first survey is views on patient feedback and the other is about the workplace culture and how person-centred it is.
  * Attend 6 x 2 hour facilitated workshops which will involve getting ready to work with patient feedback, establishing values and visions for the intervention group, critically reviewing the ways patients are offered the opportunity to give feedback
  * Engage in changes in practice (e.g. how staff offer patients the opportunity to provide feedback and the way staff make changes in response to this feedback);
  * Attend a final focus group to evaluate the workshop programme.
  Groups: Staff participants
Other: Interview — Interviews will be used to gather views about how easy or difficult it is to give feedback and how it feels to consider and/or give feedback
  Groups: Patient participants

SUMMARY:
Aim: This study aims to assess how feasible and acceptable it is to deliver facilitated team meetings, designed to support mental health teams to listen and learn from patient feedback and how helpful and feasible the evaluation methods are.

There is evidence that patients within inpatient mental health services find it difficult to share care experiences and those working in such services find it challenging to listen and act on care experience data. There is also evidence that staff burnout is higher among mental health nurses than it is in other parts of the health service.

Intervention: A team, made up of nurses, doctors, Allied Health Professionals and health care support workers working in an inpatient mental health services will engage in a 6 stage, facilitated intervention. This includes developing a more effective team culture by: getting ready for engaging with patient feedback; establishing values and vision for care experience and team work; discussing issues associated with trying to provide positive care experiences; analysis of care experiences; making change happen; reflection, evaluation and celebrating success.

Evaluation: Feasibility and acceptability will be assessed by considering views of participants and the facilitator on the intervention and ability for it to be delivered as planned. We will also consider facilitator; researcher and participants' views on the appropriateness of the evaluation methods and assess if we can achieve 50% staff response rates to a survey-person-centred practice index(PCPI). We will assess if the following methods help evaluate impact: care experiences using data from Care Opinion; complaints and feedback cards; improvement efforts made by the team in response to feedback; PCPI scores to assess changes in team culture and lastly, observations made during team meetings to assess change in team culture over time and staff survey about attitudes and beliefs about patient feedback.

DETAILED DESCRIPTION:
This study is to support health care practitioners working in acute mental health settings to build their skills and confidence in making sense of patient feedback; changing care routines; changing their ways of interacting with patients and families and with each other so that their team culture and care experience will be more person-centred.

Patient Rights (Scotland) Act 2011 requires NHS boards to listen and act on patient feedback. Previous research shows that healthcare staff working within mental health services find it challenging to listen and act on feedback. It also shows that changes they make in response to feedback tend to focus on the physical environment and not on how care is delivered or how healthcare staff behave. This study is designed to explore how these challenges can be overcome.

Some studies have, helpfully highlighted a number of factors that enhance the likelihood that teams will be able to actively engage with and act on feedback. Specifically, a number of studies have found that teams greatly benefit from facilitated support to engage effectively with feedback. There remains little understanding of what facilitation looks like or what tools are helpful in supporting learning and improving activity so if we are to become better at improving care experiences we need to urgently test interventions designed to provide such support and to evaluate them in holistic ways to understand their impact.

Health and social care services globally are exploring ways of enhancing the well-being of their workforce. NHS Grampian are committed to this and have a staff support programme, much of this current work is focused on helping people whose wellbeing has been negatively affected by work. It is necessary that we find ways in which we can support teams to be proactive about their individual and collective wellbeing which can be a protective factor against being negatively affected by team culture. Health care practitioners are also persons and as such have a need to connect with their beliefs and values. We know that health care professionals who are supported to work in ways that are consistent with their values are more likely to be able and available to offer person-centred care and are less likely to suffer from stress and burnout.

Health care practitioners working in mental health settings experience particularly high levels of distress and are often further distressed when they receive feedback that is critical of their care. The intervention, will support practitioners to address some causes of stress and burnout - namely dissatisfaction with levels of care they can provide and poor team culture and relationships.

In summary, this study works in overt ways to transform the care experiences and care and treatment of people with acute mental health, aims to enhance health care team culture and has the potential to positively impact on mental health of both patients and staff. Lastly, it may, through improvement activity that is integral to the intervention, positively impact on how services are delivered and the facilities they are delivered in."

ELIGIBILITY:
Patient inclusion criteria:

* Adults over the age of 18 who are able to give informed consent
* Current inpatient who has been admitted for at least 48 hours
* Inpatients who have been assessed by ward staff as able to participate in the study

Patient exclusion criteria

* Patients who are experiencing acute high distress and/or approach by a researcher is likely to cause more distress.
* Patients who have not been in the ward long enough (less than 48hrs) for ward staff to assess their ability to engage with the researcher.

Staff inclusion criteria

* Staff member who meets one or more of the capital criteria being used to create a team with most chance of effectively engaging and working with patient feedback (Appendix 9)
* Staff who are willing to participate in the intervention and the evaluation
* Staff whose shift pattern allow them to attend at least 80% of intervention meetings

Staff exclusion criteria:

* Staff who are unable to attend intervention delivery during the day
* Staff who are not members of the clinical or support team

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are currently inpatients within the acute mental health ward where the study is taking place.
  Staff members who work within the acute mental health ward where the study is taking place.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility | June 2023
  To understand the feasibility and acceptability of a team based intervention designed to help mental health teams listen to and act on patient experience feedback.

SECONDARY OUTCOMES:
Facilitator preparation | June 2023
  What preparation does it take for a facilitator to be able to deliver the intervention as designed?
Engagement | June 2023
  How feasible is it for a mental health team to engage with the intervention?
Acceptability | June 2023
  How acceptable is the intervention to the clinical team?
Recruitment | June 2023
  What are our recruitment rates for patients/staff participants
Time for recruitment | June 2023
  What time is required to gain recruitment of patients and staff into the study?
Methods evaluation | June 2023
  Do the methods for evaluating the impact of the intervention produce data that can be readily used to meaningfully assess the effectiveness of the intervention?
Engagement in evaluation | June 2023
  To what extent do participants engage with the evaluation methods?
Acceptability of evaluation | June 2023
  How acceptable are the methods used to evaluate the intervention to the participants?
Future sample calculation | June 2023
  Can the use of the person-centred practice index enable calculation of effect size that will enable sample calculation estimation for a future effectiveness study?

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deborah Baldie, Principal Investigator — NHS Grampian

IPD SHARING:
Plan to Share IPD: Undecided